CLINICAL TRIAL: NCT00876668
Title: Pilot-Study to Evaluate the Clinical Significance of the Fluorescence Videoangiography With Indocyanine-Green in Patients With PAD, Rutherford Classification II-V, and Relation to Common Diagnostics.
Brief Title: Evaluation of the Clinical Significance of Fluorescence Videoangiography With Indocyanine-Green
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. med. Thomas Schmitz-Rixen, Johann Wolfgang Goethe University Hospitals, Dept. of Vascular Surgery
Other Study IDs: FLAG II
Record Dates: First submitted 2008-01-16; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Peripheral Vascular Disease; Microcirculation; Ischemia
Keywords: Peripheral Vascular diseases; Microcirculation; fluorescence angiography
MeSH Terms: conditions — Peripheral Vascular Diseases; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to compare the diagnostic value of this non-invasive vascular imaging tool with the established vascular diagnostic methods for PAD in order to get prognostic data.

A higher sensitivity of Fluorescence angiography in order to recognize progression of critical limb ischemia could lead to earlier therapeutic interventions and thereby increase limb salvage. A diagnostic gap would be closed.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) occurs when the peripheral microcirculation is impaired by arterial stenoses or occlusions. In opposite to earlier studies that only evaluated intermittent claudication due to peripheral arterial disease (PAD), rest pain and trophic changes in the affected extremity are due to reduced microcirculation. Though the main reason for CLI is the existing PAD, many processes responsible for pain and other pad-associated symptoms are triggered by a reduced microcirculation so that attempts to enhance the dermal perfusion by pharmacological or other manipulations may ameliorate the results of vascular treatment. These attempts may be the best options for patients, in which vascular surgery was not successful or primarily impossible.

A Laser-induced fluorescence videoangiography is currently being used in ophthalmology to display the vessels of the eye background. Due to technical improvements, it has become a standard procedure. This trial aims at establishing laser-induced fluorescence videoangiography as standard procedure in vascular surgery. This would be of benefit for the patient as the technique does not require the use of ionising radiation and is possible for patients suffering to renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years
* Chronical ischemia of extremities, Rutherford categories 4, 5 and 6 with indication for vascular reconstruction
* Acute danger of extremity loss due tue ischemia with indication for vascular surgery

Exclusion Criteria:

* Patient < 18 years
* Informed consent not signed
* Patient has a MRSA infection
* Patient has an iodine allergy
* Pregnant female Patient
* Known anaphylactic reactions after injections of contrast media or indocyanine green

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAD, Rutherford classification II-V, not requiring surgery
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Quality of the fluorescence -videoangiography at patients with PAD | one year

SECONDARY OUTCOMES:
Correlation of the results of fluorescence videoangiography, ankle-brachial-index, i.a. DSA, clinical examination | one year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schmitz-Rixen, MD, Professor, Principal Investigator — Johann Wolfgang Goethe University Hospital

REFERENCES:
- [Background] Johnson BL, Bandyk DF, Back MR, Avino AJ, Roth SM. Intraoperative duplex monitoring of infrainguinal vein bypass procedures. J Vasc Surg. 2000 Apr;31(4):678-90. doi: 10.1067/mva.2000.104420. PMID 10753275
- [Background] Armstrong PA, Bandyk DF, Wilson JS, Shames ML, Johnson BL, Back MR. Optimizing infrainguinal arm vein bypass patency with duplex ultrasound surveillance and endovascular therapy. J Vasc Surg. 2004 Oct;40(4):724-30; discussion 730-1. doi: 10.1016/j.jvs.2004.07.037. PMID 15472601
- [Background] Heise M, Kruger U, Settmacher U, Sklenar S, Neuhaus P, Scholz H. A new method of intraoperative hydraulic impedance measurement provides valuable prognostic information about infrainguinal graft patency. J Vasc Surg. 1999 Aug;30(2):301-8. doi: 10.1016/s0741-5214(99)70141-2. PMID 10436450
- [Background] Mothes H, Donicke T, Friedel R, Simon M, Markgraf E, Bach O. Indocyanine-green fluorescence video angiography used clinically to evaluate tissue perfusion in microsurgery. J Trauma. 2004 Nov;57(5):1018-24. doi: 10.1097/01.ta.0000123041.47008.70. PMID 15580026
- [Background] Raabe A, Beck J, Gerlach R, Zimmermann M, Seifert V. Near-infrared indocyanine green video angiography: a new method for intraoperative assessment of vascular flow. Neurosurgery. 2003 Jan;52(1):132-9; discussion 139. doi: 10.1097/00006123-200301000-00017. PMID 12493110
- [Background] Holm C, Mayr M, Hofter E, Becker A, Pfeiffer UJ, Muhlbauer W. Intraoperative evaluation of skin-flap viability using laser-induced fluorescence of indocyanine green. Br J Plast Surg. 2002 Dec;55(8):635-44. doi: 10.1054/bjps.2002.3969. PMID 12550116
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Wölfle KD, Hepp W. "Intraoperative Qualitätssicherung". In: Gefäßchirurgie. Hrsg. Von Hepp W. u. Kogel. München, Jena 2000, S. 117-125